CLINICAL TRIAL: NCT01633242
Title: A Pilot Study of Cardiac Magnetic Resonance in Patients With Muscular Dystrophy
Brief Title: Heart Imaging in Children With Muscular Dystrophy
Status: Terminated | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120090; 12-H-0090
Record Dates: First submitted 2012-06-30; First posted 2012-07-04 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2016-10-11

CONDITIONS: Muscular Dystrophy
Keywords: MRI; Muscular Dystrophy; Cardiac; Myocardium; Intramyocardial fat
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Muscular dystrophy can affect the muscles used for heart function and breathing. Treatment usually involves drugs that help improve heart function. However, better types of heart imaging studies are needed to improve treatment of heart problems related to muscular dystrophy. Better heart imaging methods are especially needed for children with muscular dystrophy. Researchers want to test different heart imaging methods in children with muscular dystrophy. They will look at cardiac magnetic resonance imaging (MRI) and standard heart function tests.

Objectives:

- To develop and test new methods for imaging the heart in children with muscular dystrophy.

Eligibility:

- Children and adolescents between 8 and 17 years of age who have muscular dystrophy.

Design:

* Participants will be screened with a physical exam and medical history.
* Participants will provide a blood sample at the start of the study. They will also have heart function tests before having the imaging study.
* Participants will have a cardiac MRI scan that will last up to 60 minutes. Some tests will require a MRI contrast agent (a drug that helps the image appear more clearly on the scan).

DETAILED DESCRIPTION:
Cardiomyopathy causes significant morbidity and mortality in multiple forms of muscular dystrophy affecting children, including Duchenne muscular dystrophy (DMD), Becker muscular dystrophy (BMD) and subtypes of autosomal recessive limb-girdle muscular dystrophy (LGMD2). Pharmaceutical treatments for the cardiomyopathy of muscular dystrophy, including angiotensin-converting enzyme (ACE) inhibition and beta-adrenergic receptor blockade, afford significant benefit and demonstrate cardiac remodeling in clinical studies. Further studies are needed to identify and characterize more sensitive indicators of cardiac dysfunction in muscular dystrophy subjects to better stratify subjects for entry into clinical protocols. Using the framework of the Cooperative International Neuromuscular Research Group (CINRG) and the Clinical and Translational Science Award (CTSA) consortium, this pilot study will assess cardiac outcome measures in children obtained by gadolinium enhanced cardiac Magnetic Resonance Imaging (MRI) and echocardiographic methods that can be reliably implemented across a consortium of clinical sites devoted to the study of pharmaceutical treatments for muscular dystrophy. These cardiac MRI scans will be shared with the PITT1109 research protocol in all subjects that are enrolled in both studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or females with a diagnosis of Duchenne, Becker, or Limb Girdle Muscular Dystrophy.
* 8 to 100 years of age.

EXCLUSION CRITERIA:

* Day-time users of continuous positive airway pressure (CPAP)
* Sip ventilator users
* Invasive ventilator dependent
* Pregnant minors (when uncertain, participants will undergo urine testing) or lactating minors
* Decompensated congestive heart failure (unable to lie flat during CMR)
* Impaired renal excretory function (calculated Glomerular Filtration Rate less than 30mL/min)
* Contra-indications to Magnetic Resonance Imaging:

  * Cardiac pacemaker or implantable defibrillator
  * Cerebral aneurysm clip
  * Neural stimulator
  * Metallic ocular foreign body
  * Harrington-rod
  * Any implanted device (i.e. insulin pump, drug infusion device)
  * Claustrophobia
  * Metal shrapnel or bullet
* Investigator assessment of inability to comply with protocol
* Unable/unwilling to lie still throughout the research procedure or who require sedation
* Persons with cognitive impairment

Ages: 8 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02-24; Study Completion 2016-10-11

PRIMARY OUTCOMES:
Evaluate CMR measures in muscular dystrophy patients

SECONDARY OUTCOMES:
Early Detection
Measurement of Disease Progression
Ultimate identification of the response to developing therapies

CONTACTS AND LOCATIONS:
Overall Officials: Andrew E Arai, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hoffman EP, Brown RH Jr, Kunkel LM. Dystrophin: the protein product of the Duchenne muscular dystrophy locus. Cell. 1987 Dec 24;51(6):919-28. doi: 10.1016/0092-8674(87)90579-4. PMID 3319190
- [Background] Nigro G, Comi LI, Politano L, Bain RJ. The incidence and evolution of cardiomyopathy in Duchenne muscular dystrophy. Int J Cardiol. 1990 Mar;26(3):271-7. doi: 10.1016/0167-5273(90)90082-g. PMID 2312196
- [Background] Corrado G, Lissoni A, Beretta S, Terenghi L, Tadeo G, Foglia-Manzillo G, Tagliagambe LM, Spata M, Santarone M. Prognostic value of electrocardiograms, ventricular late potentials, ventricular arrhythmias, and left ventricular systolic dysfunction in patients with Duchenne muscular dystrophy. Am J Cardiol. 2002 Apr 1;89(7):838-41. doi: 10.1016/s0002-9149(02)02195-1. PMID 11909570